CLINICAL TRIAL: NCT02925767
Title: Efficacy of 311-nm Ti:Sapphire Laser Versus 308-nm Excimer Laser Treatment in Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jung Min Bae, Clinical Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VC16DISI0088
Record Dates: First submitted 2016-10-03; First posted 2016-10-06 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Lasers, Excimer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The 311-nm Ti:Sapphire laser treatment group (Experimental): All lesions were treated twice weekly for a total of 12-week period.
  Interventions: Device: 311-nm Ti:Sapphire laser
- The 308-nm excimer laser treatment group (Active Comparator): All lesions were treated twice weekly for a total of 12-week period.
  Interventions: Device: 308-nm excimer laser

INTERVENTIONS:
Device: 311-nm Ti:Sapphire laser — Pallas, LaserOptek, South Korea
  Arms: The 311-nm Ti:Sapphire laser treatment group
Device: 308-nm excimer laser — XTRAC, PhotoMedex, US
  Arms: The 308-nm excimer laser treatment group

SUMMARY:
A randomized controlled non-inferiority trial based on split-body was planned to compare the efficacy of 308-nm excimer laser and 311-nm Ti:Sapphire laser in patients with vitiligo.

DETAILED DESCRIPTION:
The 308-nm excimer laser (EL) has been widely used for localized vitiligo. Recently, the 311-nm Ti:Sapphire laser (TSL) was developed to treat patients with vitiligo. To compare the efficacy of TSL vs. EL in the treatment of vitiligo.

A randomized controlled non-inferiority trial based on split-body was planned. The paired symmetric vitiliginous lesions will be randomized to either TSL or EL treatment groups. All lesions will be treated twice weekly for a total of 12-week period. The degree of repigmentation will be assessed as % from baseline by using a computer program every 4 weeks, and the non-inferiority margin was set at 10%. Overall 16 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age: older than 19
* A patient with stable non-segmental vitiligo
* A patient with symmetrical vitiligo lesions
* A patient with the willingness to comply with the study protocol during the study period and capable of complying with it
* A patient who signed the informed consent prior to the participation of the study and who understands that he/she has a right to withdrawal from participation in the study at any time without any disadvantages

Exclusion Criteria:

* Age: lower than 20
* A pregnant or lactating patient
* A patient with active or spreading vitiligo
* A patient who cannot understand the study or who does not sign the informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-01-30 (Estimated); Study Completion 2018-08-30 (Estimated)

PRIMARY OUTCOMES:
The repigmentation rate (change from baseline) of the vitiliginous patch | Baseline and 12 weeks
  The degree of repigmentation will be assessed as % from baseline by using a computer program.

SECONDARY OUTCOMES:
The adverse effects of both two laser treatments | At 4 weeks, 8 weeks, and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's Hospital, Suwon, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Bae JM, Eun SH, Lee HN, Kim GM, Grimes PE, Lee JH. Comparison of 311-nm Titanium:Sapphire laser and 308-nm excimer laser treatment for vitiligo: A randomized controlled non-inferiority trial. Lasers Surg Med. 2019 Mar;51(3):239-244. doi: 10.1002/lsm.23048. Epub 2019 Jan 25. PMID 30681166